CLINICAL TRIAL: NCT04668079
Title: Comparison of Modified Cross Body Stretch and Modified Sleeper Stretch in Basketball Players for Posterior Capsule Tightness in Basketball Players
Brief Title: Modified Cross Body Stretch Verses Modified Sleeper Stretch in Basketball Players for Posterior Capsule Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00720 Rubina Naz
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Shoulder Capsulitis
Keywords: Modified cross body stretch; Modified sleeper stretch; Posterior capsule tightness; Range of motion; Seated basketball throw; Thumb up back

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified cross body stretch (Experimental): modified cross body stretch
  Interventions: Other: Modified cross body stretch
- Modified sleeper stretch (Experimental): modified sleeper stretch
  Interventions: Other: Modified sleeper stretch

INTERVENTIONS:
Other: Modified cross body stretch — Athlete was in side lying positioned. trunk was moved posteriorly 200 to 300 and shoulder is raised to 900 and semi flex both knees. Athlete was ask to passively pull the humerus across the body into horizontal adduction with the opposite hand.
  5 reps once daily 3 sets for 4 weeks was given
  Arms: Modified cross body stretch
Other: Modified sleeper stretch — Athlete was in side lying positioned on the involved side, trunk was rolled posteriorly 200 to 300 and shoulder is raised to 900 and elbow is flexed to 900 and semiflex both knees. athlete was ask to perform internal rotation passively by using the opposite arm.
  5 reps once daily 3 sets for 4 weeks was given
  Arms: Modified sleeper stretch

SUMMARY:
The aim of this research is to compare the effect of modified cross body stretch and modified sleeper stretch on pain, range of motion, disability and throwing ability in athletes with posterior capsule tightness. Randomized controlled trials done at International Islamic University. The sample size was 32. The subjects were divided in two groups, 16 subjects in modified cross body stretch group and 16 in modified sleeper stretch group. Study duration was of 6 months. Sampling technique applied was non probability connivance sampling technique. Tools used in the study are PENN shoulder score, gonoiometer, thumb up back(TUB) and seated basketball throw test(SBBT). Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Basketball is considered as the highly demanding sports due to high demand and complexity of the game. The overhead throwing activities makes it more vulnerable to the injuries. In repetitive throwing there are different type of violet forces placed on shoulder joint It causes adaptation in soft tissue anatomically which in turn limits ROM of shoulder joint and Posterior shoulder tightness.

Posterior capsule tightness can result due to abnormal humeral head motion which decreases subacromial space during overhead activities leading to compression of tissues causing limited shoulder flexion, internal rotation and horizontal adduction. Posterior capsule tightening occurs when the capsular tissue and musculature of the shoulder tighten, usually due to "repeated overload in the eccentric portion of arm deceleration. This loss of internal rotation results from contracture and tightening of the posterior inferior portion of the glenohumeral joint capsule, which occurs from the repetitive microtrauma imparted during the deceleration phase of the throwing motion. Repetitive throwing motion creates adaptive increased external rotation and decreased internal rotation in the dominant shoulder joint which is termed as GIRD (Glenohumeral internal rotation deficit).Posterior capsule tightness is often treated without surgery. It can be treated by strengthening, stretching, neuromuscular control exercises. Strengthening protocol can perform specifically on Weak muscles by using resistance and weight. The neuromuscular training helps the body to act and react on different pattern of stress demand on it through neural pathways. The mainstay of the posterior capsule tightness treatment for athlete is the stretching of the posterior capsule. One author proposed the modified forms, the modified sleeper stretch and the modified cross body stretch. And found these modified stretching more effective and beneficial than the sleeper and cross body stretch Literature review: Kevin et al investigated the acute effects of sleeper stretch on posterior shoulder tightness and internal rotation of shoulder. There was significant improvement in results.

A study conducted in 2018 to determine whether posterior shoulder stretch was effective in increasing internal rotation and horizontal adduction ROM in volleyball and tennis players with internal rotation deficit >¬¬15 degrees. The intervention group performs the sleeper stretch daily for 8 weeks. Results showed significant improvement in internal rotation and horizontal adduction.

Another article was published in 2014, with the aim to compare the effects of horizontal adduction stretch with scapular stabilization versus horizontal adduction stretch without scapular stabilization on posterior shoulder tightness and passive internal rotation. Results showed significant improvement among the scapular stabilization group.

A RCT conducted in which each subject completed stretching interventions for two days. Purpose of the study was to investigate acute effects of modified sleeper stretch and modified cross body stretch on posterior shoulder tightness and glenohumral internal rotation deficit with more than 10-degree loss.

ELIGIBILITY:
Inclusion Criteria:

* Basketball Players
* Internal rotation deficit greater than 20° degrees
* BMI 18.5-24.9

Exclusion Criteria:

* Having a systemic pathology including inflammatory joint disease
* Having musculoskeletal or neurological disease
* Having taken anti-inflammatory medication

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
PENN shoulder score | 4th week
  The disability of shoulder conditions was measured by Penn score. Which consists of 3 categories i.e.; pain, satisfaction and functional ability. Pain consists of 3 questionnaires that consists of 10 scores each (total 30) and then satisfaction, it consists of 1 questionnaire consists of 10 scores, functional ability consists of 20 questionnaires with 10 scores each for the questionnaire (total 60)
Seated basketball throw | 4th week
  SBBT (seated basketball throws) was used to test the explosiveness of the upper extremity.
Thumb up back(TUB) | 4th week
  (Thumb-up-the back- measurement) was used to measure the ability to actively move thumb up the back with the help of inch tape.

SECONDARY OUTCOMES:
Shoulder ROM (flexion) | 4th week
  Changes from the Baseline ROM range of Motion of Shoulder flexion was taken with the Help of Goniometer
Shoulder ROM Extension | 4th week
  Changes from the Baseline ROM range of Motion of Shoulder extension was taken with the Help of Goniometer
Shoulder ROM abduction | 4th week
  Changes from the Baseline ROM range of Motion of shoulder abduction was taken with the Help of Goniometer
Shoulder ROM adduction | 4th week
  Changes from the Baseline ROM range of Motion of shoulder adduction was taken with the Help of Goniometer
Shoulder ROM external rotation | 4th week
  Changes from the Baseline ROM range of Motion of Shoulder external rotation was taken with the Help of Goniometer
Shoulder ROM internal rotation | 4th week
  Changes from the Baseline ROM range of Motion of Shoulder internal rotation was taken with the Help of Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Islamic international medical college, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vukasevic V, Mitrovic M, Masanovic B. A comparative study of motor ability between elite basketball players from different regions. Sport Mont. 2020;18(1):Ahead of Print
- [Background] Ekhtiari S, Khan M, Burrus T, Madden K, Gagnier J, Rogowski JP, Maerz T, Bedi A. Hip and Groin Injuries in Professional Basketball Players: Impact on Playing Career and Quality of Life After Retirement. Sports Health. 2019 May/Jun;11(3):218-222. doi: 10.1177/1941738119838274. Epub 2019 Apr 23. PMID 31013191
- [Background] Drakos MC, Domb B, Starkey C, Callahan L, Allen AA. Injury in the national basketball association: a 17-year overview. Sports Health. 2010 Jul;2(4):284-90. doi: 10.1177/1941738109357303. PMID 23015949
- [Background] Quartey J, Davor SF, Kwakye SK. An injury profile of basketball players in Accra, Ghana. S Afr J Physiother. 2019 Mar 27;75(1):467. doi: 10.4102/sajp.v75i1.467. eCollection 2019. PMID 31061911
- [Background] Grow K. The Sleeper Stretch: Effects on Range of Motion and Injury in Baseball Players. 2010
- [Background] McClure P, Balaicuis J, Heiland D, Broersma ME, Thorndike CK, Wood A. A randomized controlled comparison of stretching procedures for posterior shoulder tightness. J Orthop Sports Phys Ther. 2007 Mar;37(3):108-14. doi: 10.2519/jospt.2007.2337. PMID 17416125
- [Background] Rao MS, Tejitha S. COMPARISON OF 3 STRETCHING PROTOCOLS FOR POSTERIOR SHOULDER TIGHTNESS IN THROWERS. Int J Physiother Res. 2016;4(2):1429-35
- [Background] Myers JB, Laudner KG, Pasquale MR, Bradley JP, Lephart SM. Glenohumeral range of motion deficits and posterior shoulder tightness in throwers with pathologic internal impingement. Am J Sports Med. 2006 Mar;34(3):385-91. doi: 10.1177/0363546505281804. Epub 2005 Nov 22. PMID 16303877
- [Background] Laudner KG, Sipes RC, Wilson JT. The acute effects of sleeper stretches on shoulder range of motion. J Athl Train. 2008 Jul-Aug;43(4):359-63. doi: 10.4085/1062-6050-43.4.359. PMID 18668168
- [Background] Chepeha JC, Magee DJ, Bouliane M, Sheps D, Beaupre L. Effectiveness of a Posterior Shoulder Stretching Program on University-Level Overhead Athletes: Randomized Controlled Trial. Clin J Sport Med. 2018 Mar;28(2):146-152. doi: 10.1097/JSM.0000000000000434. PMID 28731885
- [Background] Salamh PA, Kolber MJ, Hanney WJ. Effect of scapular stabilization during horizontal adduction stretching on passive internal rotation and posterior shoulder tightness in young women volleyball athletes: a randomized controlled trial. Arch Phys Med Rehabil. 2015 Feb;96(2):349-56. doi: 10.1016/j.apmr.2014.09.038. Epub 2014 Oct 23. PMID 25450120
- [Background] Immediate effects of two types of stretching techniques on glenohumeral internal rotation deficit and posterior shoulder tightness; a crossover randomised controlled trial